CLINICAL TRIAL: NCT01023022
Title: Medtronic CareLink® Network Evaluation Protocol
Brief Title: CareLink® Network Evaluation
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT-CareLinkEval
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2016-11

CONDITIONS: Heart Failure
Keywords: CareLink; Remote Monitoring; Cardiac Pacemaker, Artificial; Implantable Cardioverter-Defibrillators
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medtronic CareLink® Network: Patients with implanted Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy Defibrillator (CRT-D) devices, who will be monitored by the Medtronic CareLink® System.
  The System consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website.
  Interventions: Other: Medtronic CareLink® Network

INTERVENTIONS:
Other: Medtronic CareLink® Network — The Medtronic CareLink® Network consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website

SUMMARY:
The purpose of the study is to demonstrate the value of the Medtronic CareLink® Network in clinical practice in the country specific healthcare setting.

DETAILED DESCRIPTION:
Evaluation's objectives:

Comparison of remote device check and in-clinic device assessment. To assess patient ease of use of, and satisfaction with, the Medtronic CareLink® Monitor To assess clinician ease of use of, and satisfaction with, the Medtronic CareLink® Monitor and Website To assess the clinic specific clinical value of Medtronic CareLink® Network Demonstrate time savings for patients Demonstrate time savings for physicians To show the increase of efficiency through increased flexibility and per procedure time To demonstrate better handling of unscheduled activities (symptoms, events, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an implanted Medtronic ICD, CRT-D device that is supported by the Medtronic CareLink® Network
* Patients have to sign the Medtronic CareLink® "Statement of Privacy Principles" and the "Evaluation Data Protection Statement" documents

Exclusion Criteria:

* Patients with exclusion criteria required by local law
* Patient is anticipated to demonstrate poor compliance (for example, mental disturbances)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients under the care at a participating study location who have an implanted Medtronic Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy Defibrillator (CRT-D) device that is supported by the Medtronic CareLink® Network.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szwed, Prof., Principal Investigator — Institute of Cardiology, Warsaw, Poland, Spartanska 1
Locations (10):
- Poland (10):
  - I Cardiology Clinic, Clinical University Center, Gdansk
  - John Paul II Hospital, Clinic of Electrocardiology, Krakow
  - The University Hospital in Krakow; I Department of Cardiology, Krakow
  - I Department of Cardiology, Medical University in Poznan, Poznan
  - Cardiology Clinic, Pomeranian Medical University SPSK-2, Szczecin
  - Public Independent Central Clinical Hospital - SP-CSK, Warsaw
  - The Cardinal Stefan Wyszynski Institute of Cardiology, 2nd Department of Coronary Artery Disease, Warsaw
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Cardiac Arrhythmias Department, Warsaw
  - 4th Military Clinical Hospital, Clinic of Cardiology, Wroclaw
  - Silesian Medical University, Silesian Center for Heart Diseases, Clinic of Cardiology, Department of Cardiology and Inborn Defects of Heart and Electrotherapy, Zabrze

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic CareLink® Network: Patients with Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy Defibrillator (CRT-D) devices, who will be monitored by the Medtronic CareLink® System.
  The System consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website.
  Medtronic CareLink® Network: The Medtronic CareLink® Network consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website
Period: Overall Study
Arm/Group | Medtronic CareLink® Network
Started | 176 (Previous No.: 178 subjects incl. 2 pts who withdraw their approval for processing personal data)
Completed | 162
Not Completed | 14
Not completed — Death | 5
Not completed — Lost to Follow-up | 7
Not completed — due to technical issues | 2

BASELINE CHARACTERISTICS:
Groups:
- Medtronic CareLink® Network: Patients with implanted ICD or CRT-D devices, who will be monitored by the Medtronic CareLink® System.
  The System consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website.
  Medtronic CareLink® Network: The Medtronic CareLink® Network consists of the Medtronic CareLink® Monitor and Medtronic CareLink® Clinician Website
Arm/Group | Medtronic CareLink® Network
Number analyzed (Participants) | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 147
Region of Enrollment [Number; unit: participants]
  Poland | 176

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Remote Device Check and In-clinic Device Assessment
Description: "Investigators were asked the following question: how did the Medtronic CareLink system matched their personal expectation/goals and had to answer with multiple answer using the following ranking Significantly exceeded, Goals met, No expectations, Not met, Not met at all: Question 1) Newest technology for my patients. Q2) Increased patient safety. Q3) Increased patient satisfaction. Q4) Improved quality of life for my patients. Q5) Improved follow up after therapy/shock delivery of for symptomatic patients, adverse events. Q6) Increased hospital efficiency. Q7) Increased follow up quality. Q8) More flexible follow up schemes possible. Q9) Better management of the increased number of follow ups. Q10) Increased satisfaction of hospital personnel. Q11) Other goals"
Time Frame: Baseline to max. 12 months
Population: Number of Investigators who provided responded for these questions at the end of evaluation.
Measure: Number; unit: percentage of Investigators
Arm/Group | Medtronic CareLink® Network
Number analyzed (Participants) | 10
percentage of Investigators
  Answer for Qestion 1: Significantly exceeded | 40.0
  Answer for Question 1: Goals met | 50.0
  Answer for Question 1: No expectations | 10.0
  Answer for Question 1:Not met | 0.0
  Answer for Question 1:Not met at all | 0.0
  Answer for Qestion 2: Significantly exceeded | 20
  Answer for Question 2: Goals met | 80
  Answer for Question 2: No expectations | 0.0
  Answer for Question 2:Not met | 0.0
  Answer for Question 2:Not met at all | 0.0
  Answer for Qestion 3: Significantly exceeded | 10.0
  Answer for Question 3: Goals met | 70.0
  Answer for Question 3: No expectations | 20.0
  Answer for Question 3:Not met | 0.0
  Answer for Question 3:Not met at all | 0.0
  Answer for Qestion 4: Significantly exceeded | 10.0
  Answer for Question 4: Goals met | 70.0
  Answer for Question 4: No expectations | 20.0
  Answer for Question 4:Not met | 0.0
  Answer for Question 4:Not met at all | 0.0
  Answer for Qestion 5: Significantly exceeded | 30.0
  Answer for Question 5: Goals met | 70.0
  Answer for Question 5: No expectations | 0.0
  Answer for Question 5:Not met | 0.0
  Answer for Question 5:Not met at all | 0.0
  Answer for Qestion 6: Significantly exceeded | 10.0
  Answer for Question 6: Goals met | 20.0
  Answer for Question 6: No expectations | 70.0
  Answer for Question 6:Not met | 0.0
  Answer for Question 6:Not met at all | 0.0
  Answer for Qestion 7: Significantly exceeded | 10.0
  Answer for Question 7: Goals met | 60.0
  Answer for Question 7: No expectations | 30.0
  Answer for Question 7:Not met | 0.0
  Answer for Question 7:Not met at all | 0.0
  Answer for Qestion 8: Significantly exceeded | 20.0
  Answer for Question 8: Goals met | 60.0
  Answer for Question 8: No expectations | 20.0
  Answer for Question 8:Not met | 0.0
  Answer for Question 8:Not met at all | 0.0
  Answer for Qestion 9: Significantly exceeded | 20.0
  Answer for Question 9: Goals met | 60.0
  Answer for Question 9: No expectations | 20
  Answer for Question 9:Not met | 0.0
  Answer for Question 9:Not met at all | 0.0
  Answer for Qestion 10: Significantly exceeded | 10.0
  Answer for Question 10: Goals met | 20.0
  Answer for Question 10: No expectations | 50.0
  Answer for Question 10:Not met | 20.0
  Answer for Question 10:Not met at all | 0.0
  Answer for Qestion 11: Significantly exceeded | 0.0
  Answer for Question 11: Goals met | 0.0
  Answer for Question 11: No expectations | 0.0
  Answer for Question 11:Not met | 0.0
  Answer for Question 11:Not met at all | 0.0

2. Secondary Outcome: Patient Ease of Use of, and Satisfaction With the Medtronic CareLink® Monitor (Including Percentage of Patients Who Prefer Follow up With Medtronic CareLink® Compared to Traditional In-clinic Device Follow-up)
Description: "Participants were asked questions to which they could have respond multiple answers. 1) Which form of device follow up do you prefer? Answers: Monitor from home and in hospital follow up is necessary; Follow up only in hospital; No preference, and 2) How would you judge the user friendliness of the monitor in total? Answers: Very easy; Easy; Difficult; Missing Data, and 3) How did the monitor changed your daily life? did you felt more or less safe? Answers: Much more safe; Safe; No influence; Unsafe; Missing data
Time Frame: Baseline to max. 12 months
Population: Number of patients who provided responses for these questions at the end of the Study.
Measure: Number; unit: percentage of patients
Arm/Group | Medtronic CareLink® Network
Number analyzed (Participants) | 149
percentage of patients
  Question 1: Monitor f. home & in hospital f-up is | 71.8
  Question 1: Follow up only in hospital | 8.7
  Question 1: No preference | 18.8
  Question 1: Missing data | 0.7
  Question 2: Very easy | 65.1
  Question 2: Easy | 32.9
  Question 2: Difficult | 1.3
  Question 2: Missing data | 0.7
  Question 3: Much more safer | 44.3
  Question 3: Safe | 50.3
  Question 3: No influence | 4.7
  Question 3: Unsafe | 0
  Question 3: Missing data | 0.7

3. Secondary Outcome: Clinician Ease of Use of, and Satisfaction With, the Medtronic CareLink® Monitor and Website (Including Clinician General Preference, if Any, for Medtronic CareLink® Compared to Traditional In-clinic Device Follow-up)
Time Frame: Baseline to max. 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Clinic-specific Clinical Value of Medtronic CareLink® Network (Change of Workflow, Increase of Flexibility)
Time Frame: Baseline to max. 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Time and Cost Savings for Patients
Time Frame: Baseline to max. 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Time and Costs Savings for Physicians
Time Frame: Baseline to max. 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Efficiency Through Increased Flexibility and Per Procedure Time
Time Frame: Baseline to max. 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Handling of Unscheduled Activities (for Example, Symptoms and Events)
Description: "Investigators were asked to classify reasons for unscheduled visits by marking all applicable answers. Answer: 1) patient symptoms 2) adequate therapy/shock 3) appearance of already known arrythmias 4) appearance of new arrythmias 5) need for reprogramming 6) in house Follow-up 7) device alert 8) inadequate therapy/shock 9) worsening of pump function 10) malfunction of the device 11) other"
Time Frame: Baseline to max. 12 months
Population: The 68 patients of total population (176) were analyzed as this number of pt. had experienced unscheduled visit during the study.
Measure: Number; unit: % of unscheduled visits due to reasons
Units Other Than Participants: unscheduled visits
Arm/Group | Medtronic CareLink® Network
Number analyzed (Participants) | 68
Number analyzed (unscheduled visits) | 116
% of unscheduled visits due to reasons
  Reason 1: patient symptoms | 25.9
  Reason 2: adequate therapy/shock | 14.7
  Reason 3: appearance of already known arrythmias | 0.9
  Reason 4:appearance of new arrythmias | 2.6
  Reason 5: need of reprograming | 1.7
  Reason 6: in house Fup after Carelink control | 4.3
  Reason 7: device alert | 17.2
  Reason 8: inadequate therapy/shock | 6.0
  Reason 9: worsening of pump function | 0.9
  Reason 10: malfunction of the device | 0.0
  Reason 11: Other | 44.8

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only information regarding death were collected during study; none other serious and non-serious adverse events were collected.
Groups:
- Patients With Implanted ICD or CRT-D Devices: Patients with implanted ICD or CRT-D devices, who will be monitored via CareLink Network System
Arm/Group | Patients With Implanted ICD or CRT-D Devices
Serious Adverse Events (participants affected / at risk) | 5/176
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Implanted ICD or CRT-D Devices (N=176)
Death (Cardiac disorders) | 3 (3) — exacerbation of cardiac insufficiency
Death (Gastrointestinal disorders) | 1 (1) — peritonitis due to malignant sigmoid tumour
Death (General disorders) | 1 (1) — cause not determined

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less